CLINICAL TRIAL: NCT02795390
Title: Chinese and Western Medicine Collaborative Studies on Palliative Cancer Patients With Constipation
Brief Title: Clinical Trial on Palliative Cancer Patients With Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Caritas Medical Centre, Hong Kong (Other); Yan Chai Hospital (Other); Our Lady of Maryknoll Hospital (Other); Hong Kong Buddhist Hospital (Other); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Chair Professor, Director, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HKBU/KWC/PC2014
Record Dates: First submitted 2016-05-25; First posted 2016-06-10 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Constipation
Keywords: Chinese herbal medicine formula; MaZiRenWan; Randomized controlled trial; Constipation; Palliative care in cancer
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese herbal medicine (Experimental): MaZiRenWan 10g plus HuangQi 20g are chosen as the core prescription. Furthermore, six herbal granules can be added according to the syndrome differentiated for individual participant. They are ShuDiHuang 15g and Danggui 10g for deficiency of blood, Maidong 15g and ShengDiHuang 10g for deficiency of Yin, and RouCongRong 15g and Niuxi 10g for deficiency of Yang.
  Interventions: Drug: Chinese herbal medicine
- Placebo (Placebo Comparator): Placebo is made from dextrin (76.03%), tea essence (23.61%), gardenin (0.02%), and caramel (0.34%) to achieve color, smell, taste, and texture comparable to the herbal granules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chinese herbal medicine
  Arms: Chinese herbal medicine
Drug: Placebo
  Arms: Placebo

SUMMARY:
It is a double-blinded, randomized, placebo-controlled trial for advanced cancer patients with constipation. 60 patients will be randomly assigned to have individualized herbal intervention (treatment group) or placebo (control group) in 1:1 ratio. For the treatment group, MaZiRenWan 10g plus HuangQi 20g are chosen as the core prescription. Furthermore, six herbal granules can be added according to the syndrome differentiated for individual participant. Placebo is made from dextrin (76.03%), tea essence (23.61%), gardenin (0.02%), and caramel (0.34%) to achieve color, smell, taste, and texture comparable to the herbal granules. Patients are instructed to dissolve the granules in 150ml of hot water, twice daily for two weeks. The primary end point is the global symptom improvement. Secondary outcome measures include stool frequency, stool form, use of rescue herbal granules, constipation visual analogue scale (CVAS) (0=none to 7=most severe) and individual assessment of constipation related symptoms. For the safety profiles of herbal intervention, the important adverse events reported and clinical laboratory evaluations of liver and renal function are determined.

ELIGIBILITY:
Inclusion Criteria:

* Severity of constipation > 3 points (an 8-point scale from 0 to 7)
* Palliative Performance Scale ≥60%
* Relatively stable liver and renal function within 3 months
* Patients who can read and speak Chinese

Exclusion Criteria:

* Inability to communicate
* Presence of a colostomy, or gastrointestinal obstruction
* Presence of loose or watery stool (Bristol stool scale 6-7) or bowel movement > 3/day under routine laxative treatment
* History of Chinese herbal medicine allergies
* Estimated life expectancy less than 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Global symptom improvement (improved / same / worse) | 2 weeks
  Participants are asked to rate their impression of change in constipation symptoms in comparison with their baseline, with scores from 0 to 6 represents markedly worse or better at the respective extremes. The response categories are collapsed to simply "improved" for score 4-6, "same" for score 3, or "worse" for score 0-2.

SECONDARY OUTCOMES:
Number of bowel movement (times/day) | 2 weeks
Stool form | 2 weeks
  Stool form is assessed with 7-point Bristol Stool Scale (ranging from "separate hard lumps" to "watery")
Extra laxatives used (times/week) | 2 week
Constipation visual analogue scale | 2 weeks
  The severity of constipation is evaluated by an eight point ordinal rating scale (0=none to 7=most severe)
Constipation related symptoms | 2 weeks
  Sensation of straining, incomplete evacuation, bloating, abdominal pain/cramping, nausea, and passing of gas are recorded using a 7-point ordinal scale (0=not at all and 6=very severe)
Adverse events | 2 weeks
Blood creatinine level (umol/L) | 2 weeks
Blood urea level (mmol/L) | 2 weeks
Serum glutamic pyruvic transaminase(SGPT) Level (U/L) | 2 weeks
Serum Glutamic Oxaloacetic Transaminase (SGOT) Level (U/L) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-xiang Bian, PhD, Principal Investigator — Hong Kong Baptist University
Locations (3):
- Hong Kong (3):
  - Caritas Medical Centre, Hong Kong
  - Hong Kong Buddhist Hospital, Hong Kong
  - Our Lady of Maryknoll Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research results will be published after analysis.
Supporting Information: Study Protocol, ICF
Time Frame: After publication with no time limit
Access Criteria: Open for public

REFERENCES:
- [Derived] Cheng CW, Mok HF, Yau CWS, Chan JTM, Kang YC, Lam PY, Zhong LLD, Zhao C, Ng BFL, Kwok AOL, Tse DMW, Bian ZX. A pilot randomized placebo-controlled study on modified MaZiRenWan: a formulated Chinese medicine to relieve constipation for palliative cancer patients. Chin Med. 2022 Mar 2;17(1):31. doi: 10.1186/s13020-022-00580-0. PMID 35236375